CLINICAL TRIAL: NCT03460028
Title: Evaluation of the Transitional Pain Service Surgical Oncology Yoga Program for Individuals With Persistent Pain; a Pilot Randomized Controlled Trial
Brief Title: Yoga for Persistent Pain Related to Oncology Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-5942.0
Record Dates: First submitted 2017-10-17; First posted 2018-03-09 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Persistent Postoperative Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Condition (Experimental): Participants randomized to the Yoga Condition will participate in a specialized yoga intervention.
  Interventions: Behavioral: Yoga Condition
- Wait-List Control Condition (No Intervention): Participants randomized to the Wait-List Control Condition will participate in a specialized yoga intervention once the Yoga Condition has completed their assigned intervention.

INTERVENTIONS:
Behavioral: Yoga Condition — Participants randomized to the Yoga Condition will participate in an integrated yoga program consisting of yoga postures, breathing exercises, and concentration/meditation practices.
  Arms: Yoga Condition

SUMMARY:
This randomized controlled trial will evaluate a yoga intervention for individuals who experience persistent pain following oncology surgery. The integrated yoga program will involve postures, breathing exercises, and concentration practices. Data will be collected at several time points (pre-, mid-, and post-intervention) for both the intervention and wait-list control conditions. The data will be analysed using linear mixed effects growth models. Results will be written up in manuscript format, published in a peer review journal, and disseminated at scientific research conferences.

ELIGIBILITY:
Inclusion Criteria:

1. Is a patient at specific pain clinics
2. Has undergone oncology surgery prior to commencing the yoga intervention
3. Is 18 years of age or older
4. Is able to speak and read English
5. Is able to commit to one weekly, one hour yoga classes for eight weeks
6. Is able to provide a note from their physician or kinesiologist indicating that it is safe for them to participate in a gentle physical activity intervention, such as yoga

Exclusion Criteria:

1. Has pre-existing medical contraindications that preclude participation
2. Has cognitive limitations or language comprehension issues that would impact participation
3. Have had a regular yoga practice in the last six months
4. Documented personality disorder
5. Pregnant women
6. Current enrollment in another research trial evaluating a mind-body intervention

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in scores on the Pain Catastrophizing Scale | at 0, 4 and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada